CLINICAL TRIAL: NCT02975102
Title: A Study to Evaluate the Performance and Safety of CBL-101 Versus Vismed® Multi Eye Drops in the Management of Dry Eye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoire Chauvin (Industry)
Collaborators: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-A01121-50
Record Dates: First submitted 2016-11-21; First posted 2016-11-29 (Estimated); Results first posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-01

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBL-101 Eye Drops (Experimental): The test article, CBL-101 Eye Drops, is a CE-marked medical device containing 0.15% sodium hyaluronate and polyethylene glycol (PEG) 8000. An oxide (Oxyd®) used as a soft preservative, rapidly turns into oxygen, water and ions on contact with the eye. The formula is presented in 10 mL bottles.
  Interventions: Device: CBL-101 Eye Drops
- Vismed® Multi Eye Drops (Active Comparator): The comparator product, Vismed® Multi ophthalmic solution (CE marked), contains 0.18% sodium hyaluronate, is unpreserved and presented in 10 mL bottles.
  Interventions: Device: Vismed® Multi Eye Drops

INTERVENTIONS:
Device: CBL-101 Eye Drops — CBL-101 Eye Drops 3 to 6 times per day for 3 months.
  Arms: CBL-101 Eye Drops
Device: Vismed® Multi Eye Drops — Vismed® Multi 3 to 6 times per day for 3 months.
  Arms: Vismed® Multi Eye Drops

SUMMARY:
The primary objectives of this investigation are to show that the performance of CBL-101 Eye Drops is non-inferior to that of Vismed® Multi eye drops in subjects with moderate to severe keratoconjunctivitis sicca after 28 days, and to assess the safety of CBL-101 Eye Drops during a 90-day period with treatment administered 3 to 6 times per day.

DETAILED DESCRIPTION:
Participants in this multicenter, randomized study had a screening visit, then were randomized on Day 0 with follow-up visits on Day 7 (±1), Day 28 (± 3) and Day 90 (±10).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be of legal age (at least 18) on the date the Informed Consent Form (ICF) is signed and with the capacity to provide voluntary informed consent
2. Subjects must be able to read, understand, and provide written informed consent on the Ethics Committee (EC) approved ICF
3. Subjects who are able and willing to comply with all treatment and follow-up, study procedures
4. Subjects who have been using tear substitutes for at least 3 months prior to inclusion, and who will use multidose preservative-free artificial tear (Aqualarm U.P. povidone 2% eye drops in 10 mL bottles) up to 6 times a day for at least 2 weeks immediately prior to randomization
5. Subjects with a score ≥ 1 for at least 2 out of the 7 following symptoms (rated 0 to 4): sensation of dryness, foreign body, burning, stinging, itching, blurred vision, sensitivity to light
6. Subjects with at least 1 eye with the following signs of keratoconjunctivitis sicca :

   * Tear break-up time of ≤ 10sec (mean of 3 measurements) at both screening visit and inclusion visit
   * Total ocular surface staining score ≥ 4 and ≤ 9 at both screening visit and inclusion visit. This assessment combines corneal, nasal and temporal bulbar conjunctival fluorescein staining, each graded 0-5 according to the Oxford Scheme
7. Subjects who have a decimal visual acuity (VA) with habitual correction equal to or better than 0.1 (Monoyer chart) in both eyes
8. Subjects with no systemic treatment or who are receiving stable systemic treatment (unchanged for 1 month or longer)
9. Female subjects who are not of childbearing potential or who have a negative urine pregnancy test result at screening

Exclusion Criteria:

Ocular Exclusion Criteria

1. Subjects with moderate or severe blepharitis defined by at least moderate (a score of ≥ 2 from a range of 0 to 3) eyelid margin hyperemia or moderate eyelid swelling or both and at least moderate eyelid debris or moderate plugging of meibomian glands or both
2. Subjects who have severe ocular dryness accompanied by one of the following:

   * Lid abnormality (except mild blepharitis)
   * Corneal disease
   * Ocular surface metaplasia
   * Filamentary keratitis
   * Corneal neovascularization
3. Subjects who currently wear contact lenses or have worn contact lenses within 90 days prior to study start
4. Subjects who have received ocular surgery, including laser surgery, in either eye within 180 days prior to study start
5. Subjects with a history of ocular trauma, non-dry eye ocular inflammation, or ocular infection within 90 days prior to study start
6. Subjects with a history of ocular allergic disease or ocular herpes within 1 year prior to study start
7. Subjects with a history of any inflammatory ulcerative keratitis, recurrent corneal erosion, or uveitis

   Treatment Exclusion Criteria
8. Subjects with known hypersensitivity or contraindications to any of the ingredients in the test or comparator products or ART
9. Subjects with initiation of, or changes to, concomitant medication that could affect dry eye within 30 days prior to Visit 1 (Screening) or with planned initiation or changes of such medications during the study
10. Subjects who have received ocular therapy (either eye) with any ophthalmic medication, except tear substitutes, within 2 weeks prior to study start
11. Subjects expected to receive ocular therapy during the study
12. Subjects treated with topical ocular steroidal or non-steroidal antiinflammatory medication within 30 days prior to study start
13. Subjects expected to receive ocular therapy with immunosuppressants (e.g. cyclosporine) during the study or who have used ocular immunosuppressants within 90 days prior to study start
14. Subjects who have received occlusion therapy with lacrimal or punctum plugs within 90 days prior to study start

    General Exclusion Criteria
15. Female subjects who are sexually active and who do not fall into 1 of the following categories:

    * Post-menopausal
    * Surgically sterile
    * Using one of the following birth control methods throughout the duration of the study: Intrauterine device (at least for 14 days prior to study start) or Barrier method (condom or diaphragm) with spermicide (at least for 14 days prior to study start) or Hormonal contraception (same dose and same formulation for at least 6 months)
16. Females who are breastfeeding
17. Subjects participating in any drug or device clinical investigation within 30 days prior to entry into this study and, or during the period of study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raphaele Siou Mermet, MD, Study Director — Laboratoire Chauvin
Locations (2):
- Dr. Nyst private office, Huy, Belgium
- Pr Mortemousque private office, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Labetoulle M, Mortemousque B; CBL-101 Study Group. Performance and Safety of a Sodium Hyaluronate Tear Substitute with Polyethylene Glycol in Dry Eye Disease: A Multicenter, Investigator-Masked, Randomized, Noninferiority Trial. J Ocul Pharmacol Ther. 2022 Nov;38(9):607-616. doi: 10.1089/jop.2022.0048. Epub 2022 Oct 21. PMID 36269661

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 15 sites in France and 3 sites in Belgium
Pre-assignment Details: 87 enrolled participants underwent a washout period of 2 weeks with povidone 2% eye drops in both eyes. Following completion of the washout period, 83 participants met inclusion criteria and were randomized either to CBL-101 or Vismed Multi treatment group. Both eyes of each participant were treated with the assigned eye drops.
Groups:
- CBL-101 Eye Drops: Participants received CBL-101 Eye Drops, 3 to 6 times daily for 3 months in both eyes.
  CBL-101 Eye Drops: CE-marked medical device with 0.15% sodium hyaluronate and 0.5% polyethylene glycol (PEG)
- Vismed® Multi Eye Drops: Participants received Vismed® Multi Eye Drops, 3 to 6 times daily for 3 months in both eyes.
  Vismed® Multi: CE-marked medical device with 0.18% sodium hyaluronate
Period: Overall Study
Arm/Group | CBL-101 Eye Drops | Vismed® Multi Eye Drops
Started (Randomized) | 45 | 38
Safety Population | 45 | 38
Intention-to-treat Population | 45 | 38
Per Protocol Population Day 7 | 42 (One participant did not attend the Day 7 visit. 2 participants were excluded for major deviation: 1 withdrawal before Day 28, 1 had disallowed concomitant therapy.) | 34 (One participant did not attend the Day 7 visit. 3 participants were excluded for major deviation:3 had inclusion criteria violation.)
Per Protocol Population Day 28 | 43 (2 participants were excluded for major deviation: 1 withdrawal before Day 28, 1 had disallowed concomitant therapy) | 35 (3 participants were excluded for major deviation:3 had inclusion criteria violation)
Per Protocol Population Day 90 | 42 (One participant withdrew after Day 28) | 34 (One participant withdrew after Day 28)
Completed | 43 | 37
Not Completed | 2 | 1
Not completed — Adverse Event | 2 | 1

BASELINE CHARACTERISTICS:
Population: Baseline participants included all 83 randomized participants.
Groups:
- CBL-101 Eye Drops: Participants received CBL-101 Eye Drops, 3 to 6 times daily for 3 months in both eyes.
  CBL-101 Eye Drops: CE-marked medical device with 0.15% sodium hyaluronate, and 0.5% polyethylene glycol (PEG)
- Total: Total of all reporting groups
Arm/Group | CBL-101 Eye Drops | Vismed® Multi Eye Drops | Total
Number analyzed (Participants) | 45 | 38 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (14.0) | 60.6 (14.1) | 62.3 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 29 | 63
  Male | 11 | 9 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 39 | 33 | 72
  Belgium | 6 | 5 | 11
Ocular surface fluorescein staining [Mean (Standard Deviation); unit: units on a scale] — The Ocular Surface Fluorescein Staining (OSFS) was scored according to a scale (Oxford Scheme) with a total score ranging from a minimum of 0 (best outcome) to a maximum of 15 (worst outcome).
  The OSFS total score is the sum of 3 subscores (corneal, nasal and temporal regions). Each subscore ranges from a minimum of 0 (best outcome) to a maximum of 5 (worst outcome).
  units on a scale | 5.4 (1.3) | 5.3 (1.5) | 5.3 (1.4)
Corneal fluorescein staining score [Mean (Standard Deviation); unit: units on a scale] — The Corneal fluorescein staining score was measured according to a scale (Oxford Scheme) ranging from a minimum of 0 (best outcome) to a maximum of 5 (worst outcome).
  units on a scale | 1.8 (0.7) | 1.9 (0.8) | 1.9 (0.8)
Nasal conjunctival fluorescein staining score [Mean (Standard Deviation); unit: units on a scale] — The Nasal conjunctival fluorescein staining score was measured according to a scale (Oxford Scheme) ranging from a minimum of 0 (best outcome) to a maximum of 5 (worst outcome).
  units on a scale | 1.8 (0.7) | 1.7 (0.7) | 1.8 (0.7)
Temporal conjunctival fluorescein staining score [Mean (Standard Deviation); unit: units on a scale] — The Temporal conjunctival fluorescein staining score was measured according to a scale (Oxford Scheme) ranging from a minimum of 0 (best outcome) to a maximum of 5 (worst outcome).
  units on a scale | 1.7 (0.7) | 1.7 (0.5) | 1.7 (0.6)
Global dry eye symptoms score [Mean (Standard Deviation); unit: units on a scale] — The Global dry eye symptom score was the sum score (scale 0-28) of dry eye symptoms assessing 7 items: sensation of dryness, foreign body, burning, stinging, itching, blurred vision, sensitivity to light, each graded from 0 (absent) to 4 (severe and/or disabling and constant).
  units on a scale | 8.8 (2.7) | 8.2 (3.3) | 8.5 (3.0)
Ocular surface disease-Quality of life (OSD-QoL®): Global question [Mean (Standard Deviation); unit: units on a scale] — The Global Question of the OSD-QoL questionnaire was measured on a scale ranging from 0 (worst outcome) to 4 (best outcome). The result was converted to a reporting score ranging from 0 (poor quality of life) to 100 (good quality of life). Population: Some of the Quality of Life questionnaires could not be analyzed
  units on a scale
    number analyzed (Participants) | 40 | 32 | 72
    (all) | 45.6 (21.8) | 53.9 (22.1) | 49.3 (22.2)
Tear film break-up time (TFBUT) [Mean (Standard Deviation); unit: seconds] — The Tear Film Break Up Time (TFBUT) after fluorescein instillation, measured the time between the last blink and the first appearance of a dry spot or disruption of the tear film. The TFBUT was measured in tenths of seconds with a stopwatch provided to the sites. It was conducted 3 times and the mean was calculated.
  seconds | 5.5 (1.6) | 6.0 (1.5) | 5.7 (1.6)
Schirmer's test [Mean (Standard Deviation); unit: millimeters] — Tear fluid secretion was assessed by the unanaesthetized Schirmer's test in the study eye with graduated strips in millimeters.
  Schirmer paper test strips were carefully inserted over the lower eyelid margin. The strips were removed after 5 minutes and the amount of tear fluid secretion read to the nearest mm from the graduated strip markings.
  millimeters | 6.8 (3.7) | 7.4 (2.9) | 7.1 (3.3)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Ocular Surface Fluorescein Staining Score at Day 28
Description: Mean change from baseline (CFB) in the study eye in Ocular Surface Fluorescein Staining (OSFS) scored according to the Oxford Scheme.
  The Oxford Scheme is a validated scale consisting of a series of panels labelled A to E in order of increasing severity. Grade 0 corresponds to panel A increasing to Grade 5 corresponding to more than Panel E, with punctate dots representing staining. The 3 regions, cornea, nasal and temporal bulbar conjunctiva are graded separately from 0 to 5, with the OSFS score ranging from 0 (best outcome) to 15 (worst outcome). The OSFS is the sum score of the 3 subscores (cornea, nasal and temporal regions).
  The study eye was the eligible eye with the highest OSFS score at baseline, which needed to be ≥4 and ≤9 on the 15-grade Oxford Scheme. If both eyes were eligible and had the same OSFS score, the study eye was the right eye.
Time Frame: Baseline (Day 0), Visit 4 (Day 28)
Population: Analysis was performed as planned on the Per-protocol population (78 participants) . The Per-protocol population consisted of all randomized participants with at least one instillation and one post-baseline assessment without any major protocol deviation (defined as impacting the primary endpoint)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CBL-101 Eye Drops | Vismed® Multi Eye Drops
Number analyzed (Participants) | 43 | 35
score on a scale | -2.9 (0.3) | -2.4 (0.3)
Statistical Analysis 1: Comparison: CBL-101 Eye Drops vs Vismed® Multi Eye Drops; Test type: Non-Inferiority — A sample size of 33 evaluable patients per treatment group was calculated to provide at least 90% power to demonstrate non-inferiority of CBL-101 to Vismed Multi. Assumptions included a non-inferiority margin of 2 grades and a standard deviation of 2.5; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-1.2 to 0.3], Standard Error of Mean 0.4 — Treatment difference : CBL-101 - Vismed Multi

2. Secondary Outcome: Change From Baseline in Ocular Surface Fluorescein Staining Score at Day 7 (Visit 3)
Description: as for outcome 1
Time Frame: Baseline (Day 0), Visit 3 (Day 7)
Population: Analysis was performed on the Per-protocol population as planned. Two participants of the per-protocol population, one in each group did not have the Day 7 visit.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CBL-101 Eye Drops | Vismed® Multi Eye Drops
Number analyzed (Participants) | 42 | 34
score on a scale | -1.7 (0.2) | -1.4 (0.2)
Statistical Analysis 1: Comparison: CBL-101 Eye Drops vs Vismed® Multi Eye Drops; Test type: Superiority; p > 0.05, ANCOVA — Significance level of 0.05; Adjustment for baseline

3. Secondary Outcome: Change From Baseline in Ocular Surface Fluorescein Staining Score at Day 90 (Visit 5)
Description: as for outcome 1
Time Frame: Baseline (Day 0), Visit 5 (Day 90)
Population: Two participants of the per-protocol population, one in each group withdrew before the Day 90 visit.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CBL-101 Eye Drops | Vismed® Multi Eye Drops
Number analyzed (Participants) | 42 | 34
score on a scale | -4.0 (0.2) | -2.6 (0.3)
Statistical Analysis 1: Comparison: CBL-101 Eye Drops vs Vismed® Multi Eye Drops; Test type: Superiority; p = 0.0002, ANCOVA — Significance level of 0.05; Adjustment for baseline

4. Secondary Outcome: Change From Baseline in Corneal Fluorescein Staining Score at Day 7 (Visit 3)
Description: Mean change from baseline (CFB) in the study eye in Corneal Fluorescein Staining scored according to the Oxford Scheme.
  The Oxford Scheme is a validated scale consisting of a series of panels labelled A to E in order of increasing severity. Grade 0 corresponds to panel A increasing to Grade 5 corresponding to more than Panel E, with punctate dots representing staining. The Corneal region is graded separately from 0 (best outcome) to 5 (worst outcome).
Time Frame: Baseline (Day 0), Visit 3 (Day 7)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CBL-101 Eye Drops | Vismed® Multi Eye Drops
Number analyzed (Participants) | 42 | 34
score on a scale | -0.5 (0.1) | -0.4 (0.1)
Statistical Analysis 1: Comparison: CBL-101 Eye Drops vs Vismed® Multi Eye Drops; Test type: Superiority; p > 0.05, ANCOVA — Significance level of 0.05; Adjustment for baseline

5. Secondary Outcome: Change From Baseline in Corneal Fluorescein Staining Score at Day 28 (Visit 4)
Description: as for outcome 4
Time Frame: Baseline (Day 0), Visit 4 (Day 28)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CBL-101 Eye Drops | Vismed® Multi Eye Drops
Number analyzed (Participants) | 43 | 35
score on a scale | -0.9 (0.1) | -0.8 (0.1)
Statistical Analysis 1: Comparison: CBL-101 Eye Drops vs Vismed® Multi Eye Drops; Test type: Superiority; p > 0.05, ANCOVA — Significance level of 0.05; Adjustment for baseline

6. Secondary Outcome: Change From Baseline in Corneal Fluorescein Staining Score at Day 90 (Visit 5)
Description: as for outcome 4
Time Frame: Baseline (Day 0), Visit 5 (Day 90)
Population: Two participants of the per-protocol population, one in each group withdrew before the Day 90 visit.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CBL-101 Eye Drops | Vismed® Multi Eye Drops
Number analyzed (Participants) | 42 | 34
score on a scale | -1.2 (0.1) | -0.8 (0.1)
Statistical Analysis 1: Comparison: CBL-101 Eye Drops vs Vismed® Multi Eye Drops; Test type: Superiority; p = 0.0186, ANCOVA — Significance level of 0.05; Adjustment for baseline

7. Secondary Outcome: Change From Baseline in Nasal Conjunctival Fluorescein Staining Score at Day 7 (Visit 3)
Description: Mean change from baseline (CFB) in the study eye in Nasal conjunctival Fluorescein Staining scored according to the Oxford Scheme.
  The Oxford Scheme is a validated scale consisting of a series of panels labelled A to E in order of increasing severity. Grade 0 corresponds to panel A increasing to Grade 5 corresponding to more than Panel E, with punctate dots representing staining. The Nasal conjunctival region is graded separately from 0 (best outcome) to 5 (worst outcome).
Time Frame: Baseline (Day 0), Visit 3 (Day 7)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CBL-101 Eye Drops | Vismed® Multi Eye Drops
Number analyzed (Participants) | 42 | 34
score on a scale | -0.6 (0.1) | -0.6 (0.1)
Statistical Analysis 1: Comparison: CBL-101 Eye Drops vs Vismed® Multi Eye Drops; Test type: Superiority; p > 0.05, ANCOVA — Significance level of 0.05; Adjustment for baseline

8. Secondary Outcome: Change From Baseline in Nasal Conjunctival Fluorescein Staining Score at Day 28 (Visit 4)
Description: as for outcome 7
Time Frame: Baseline (Day 0), Visit 4 (Day 28)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CBL-101 Eye Drops | Vismed® Multi Eye Drops
Number analyzed (Participants) | 43 | 35
score on a scale | -1.0 (0.1) | -0.9 (0.1)
Statistical Analysis 1: Comparison: CBL-101 Eye Drops vs Vismed® Multi Eye Drops; Test type: Superiority; p > 0.05, ANCOVA — Significance level of 0.05; Adjustment for baseline

9. Secondary Outcome: Change From Baseline in Nasal Conjunctival Fluorescein Staining Score at Day 90 (Visit 5)
Description: as for outcome 7
Time Frame: Baseline (Day 0), Visit 5 (Day 90)
Population: Two participants of the per-protocol population, one in each group withdrew before the Day 90 visit.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CBL-101 Eye Drops | Vismed® Multi Eye Drops
Number analyzed (Participants) | 42 | 34
score on a scale | -1.4 (0.1) | -0.8 (0.1)
Statistical Analysis 1: Comparison: CBL-101 Eye Drops vs Vismed® Multi Eye Drops; Test type: Superiority; p = 0.0011, ANCOVA — Significance level of 0.05; Adjustment for baseline

10. Secondary Outcome: Change From Baseline in Temporal Conjunctival Fluorescein Staining Score at Day 7 (Visit 3)
Description: Mean change from baseline (CFB) in the study eye in Temporal Conjunctival Fluorescein Staining scored according to the Oxford Scheme.
  The Oxford Scheme is a validated scale consisting of a series of panels labelled A to E in order of increasing severity. Grade 0 corresponds to panel A increasing to Grade 5 corresponding to more than Panel E, with punctate dots representing staining. The Temporal conjunctival region is graded separately from 0 (best outcome) to 5 (worst outcome).
Time Frame: Baseline (Day 0), Visit 3 (Day 7)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CBL-101 Eye Drops | Vismed® Multi Eye Drops
Number analyzed (Participants) | 42 | 34
score on a scale | -0.6 (0.1) | -0.4 (0.1)
Statistical Analysis 1: Comparison: CBL-101 Eye Drops vs Vismed® Multi Eye Drops; Test type: Superiority; p > 0.05, ANCOVA — Significance level of 0.05; Adjustment for baseline

11. Secondary Outcome: Change From Baseline in Temporal Conjunctival Fluorescein Staining Score at Day 28 (Visit 4)
Description: as for outcome 10
Time Frame: Baseline (Day 0), Visit 4 (Day 28)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CBL-101 Eye Drops | Vismed® Multi Eye Drops
Number analyzed (Participants) | 43 | 35
score on a scale | -0.9 (0.1) | -0.8 (0.1)
Statistical Analysis 1: Comparison: CBL-101 Eye Drops vs Vismed® Multi Eye Drops; Test type: Superiority; p > 0.05, ANCOVA — Significance level of 0.05; Adjustment for baseline

12. Secondary Outcome: Change From Baseline in Temporal Conjunctival Fluorescein Staining Score at Day 90 (Visit 5)
Description: as for outcome 10
Time Frame: Baseline (Day 0), Visit 5 (Day 90)
Population: Two participants of the per-protocol population, one in each group withdrew before the Day 90 visit.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CBL-101 Eye Drops | Vismed® Multi Eye Drops
Number analyzed (Participants) | 42 | 34
score on a scale | -1.4 (0.1) | -0.9 (0.1)
Statistical Analysis 1: Comparison: CBL-101 Eye Drops vs Vismed® Multi Eye Drops; Test type: Superiority; p = 0.005, ANCOVA — Significance level of 0.05; Adjustment for baseline

13. Secondary Outcome: Change From Baseline in Global Sum Score of Dry Eye Symptoms at Day 28 (Visit 4)
Description: The global sum score (scale 0-28) of dry eye symptoms assessed 7 items: sensation of dryness, foreign body, burning, stinging, itching, blurred vision, sensitivity to light, each graded from 0 (absent) to 4(severe and/or disabling and constant).
Time Frame: Baseline, Visit 4 (Day 28)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CBL-101 Eye Drops | Vismed® Multi Eye Drops
Number analyzed (Participants) | 43 | 35
score on a scale | -4.2 (0.4) | -2.2 (0.4)
Statistical Analysis 1: Comparison: CBL-101 Eye Drops vs Vismed® Multi Eye Drops; Test type: Superiority; p = 0.0008, ANCOVA — Significance level of 0.05; Adjustment for baseline

14. Secondary Outcome: Change From Baseline in Global Sum Score of Dry Eye Symptoms at Day 90 (Visit 5)
Description: The global sum score (scale 0-28) of dry eye symptoms assessed 7 items: sensation of dryness, foreign body, burning, stinging, itching, blurred vision, sensitivity to light, each graded from 0 (absent) to 4 (severe and/or disabling and constant).
Time Frame: Baseline, Visit 5 (Day 90)
Population: Two participants of the per-protocol population, one in each group withdrew before the Day 90 visit.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CBL-101 Eye Drops | Vismed® Multi Eye Drops
Number analyzed (Participants) | 42 | 34
score on a scale | -5.1 (0.4) | -3.1 (0.5)
Statistical Analysis 1: Comparison: CBL-101 Eye Drops vs Vismed® Multi Eye Drops; Test type: Superiority; p = 0.0026, ANCOVA — Significance level of 0.05; Adjustment for baseline

15. Secondary Outcome: Change From Baseline in the Ocular Surface Disease-Quality of Life (OSD-QoL®) at Day 90 (Visit 5)
Description: The OSD-QoL® questionnaire is a validated instrument for measuring dry eye severity and impairment. It includes 28 items divided into 7 dimensions: Daily activities, Difficulties with work and handicap, Giving up makeup, Acknowledgement of the disease, Acceptance of the disease, Fear for the future, and Emotional well-being. A Global Question: "How do you feel when considering your eye problems?" (included in the Fear for the future dimension) was also evaluated separately. The converted score for each dimension ranges from 0 to 100, with a higher score reflecting a better quality of life.
Time Frame: Baseline (Day 0), Visit 5 (Day 90)
Population: Analysis population included participants in the per-protocol population with evaluable Global question on Day 0 and Day 90.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CBL-101 Eye Drops | Vismed® Multi Eye Drops
Number analyzed (Participants) | 37 | 28
score on a scale
  Daily activities: number analyzed (Participants) | 37 | 27
  Daily activities | 12.0 (1.9) | 5.3 (2.2)
  Handicap and work difficulties: number analyzed (Participants) | 23 | 24
  Handicap and work difficulties | 10.8 (2.0) | 2.4 (2.0)
  Giving up makeup: number analyzed (Participants) | 25 | 22
  Giving up makeup | 12.2 (3.9) | 5.5 (4.2)
  Acknowledgement of the disease | 5.8 (3.6) | 2.6 (4.2)
  Acceptance of the disease | 0.5 (3.6) | -1.5 (4.1)
  Fear for the future | 15.5 (2.2) | 5.3 (2.6)
  Emotional well-being: number analyzed (Participants) | 36 | 27
  Emotional well-being | 6.8 (1.9) | 2.6 (2.2)
  Global Question | 17.5 (3.0) | 9.1 (3.5)
Statistical Analysis 1: Comparison: CBL-101 Eye Drops vs Vismed® Multi Eye Drops; Test type: Superiority; p = 0.077, ANCOVA — Significance level of 0.05 . P-Value result provided only for Global Question; Adjustment for baseline

16. Secondary Outcome: Change From Baseline in Tear Film Break Up Time (TFBUT) at Day 7 (Visit 3)
Description: The Tear Film Break Up Time (TFBUT) after fluorescein instillation, measured the time between the last blink and the first appearance of a dry spot or disruption of the tear film. The TFBUT was measured in tenths of seconds with a stopwatch provided to the sites. It was conducted 3 times and the mean was calculated.
Time Frame: Baseline (Day 0), Visit 3 (Day 7)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | CBL-101 Eye Drops | Vismed® Multi Eye Drops
Number analyzed (Participants) | 42 | 34
seconds | 0.9 (0.2) | 0.7 (0.2)
Statistical Analysis 1: Comparison: CBL-101 Eye Drops vs Vismed® Multi Eye Drops; Test type: Superiority; p = 0.6097, ANCOVA — Significance level of 0.05; Adjustment for baseline

17. Secondary Outcome: Change From Baseline in Tear Film Break Up Time (TFBUT) at Day 28 (Visit 4)
Description: The Tear Film Break Up Time (TFBUT) after fluorescein instillation, measured the time between the last blink and the first appearance of a dry spot or disruption of the tear film. The TFBUT was measured in tenths of seconds with a stopwatch provided to the sites. It was conducted 3 times and the means was calculated.
Time Frame: Baseline (Day 0), Visit 4 (Day 28)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | CBL-101 Eye Drops | Vismed® Multi Eye Drops
Number analyzed (Participants) | 43 | 35
seconds | 1.2 (0.2) | 0.8 (0.2)
Statistical Analysis 1: Comparison: CBL-101 Eye Drops vs Vismed® Multi Eye Drops; Test type: Superiority; p = 0.231, ANCOVA — Significance level of 0.05; Adjustment for baseline

18. Secondary Outcome: Change From Baseline in Tear Film Break Up Time (TFBUT) at Day 90 (Visit 5)
Description: as for outcome 17
Time Frame: Baseline (Day 0), Visit 5 (Day 90)
Population: Two participants of the per-protocol population, one in each group withdrew before the Day 90 visit.
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | CBL-101 Eye Drops | Vismed® Multi Eye Drops
Number analyzed (Participants) | 42 | 34
seconds | 1.7 (0.2) | 0.7 (0.3)
Statistical Analysis 1: Comparison: CBL-101 Eye Drops vs Vismed® Multi Eye Drops; Test type: Superiority; p = 0.0135, ANCOVA — Significance level of 0.05; Adjustment for baseline

19. Secondary Outcome: Change From Baseline in Schirmer Test at Day 28 (Visit 4)
Description: Tear fluid secretion was assessed by the unanaesthetized Schirmer's test in the study eye with graduated strips in millimeters.
  Schirmer paper test strips were carefully inserted over the lower eyelid margin. The strips were removed after 5 minutes and the amount of tear fluid secretion read to the nearest mm from the graduated strip markings.
Time Frame: Baseline (Day 0), Visit 4 (Day 28)
Population: Analysis population included participants in the per-protocol population with evaluable Schirmer test on Day 0 and Day 28.
Measure: Least Squares Mean (Standard Error); unit: mm / 5 min
Arm/Group | CBL-101 Eye Drops | Vismed® Multi Eye Drops
Number analyzed (Participants) | 41 | 34
mm / 5 min | 1.9 (0.5) | 1.5 (0.5)
Statistical Analysis 1: Comparison: CBL-101 Eye Drops vs Vismed® Multi Eye Drops; Test type: Superiority; p = 0.575, ANCOVA — Significance level of 0.05; Adjustment for baseline

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the whole treatment period from the first instillation until the last study visit (90 ± 10 days).
Description: Any untoward medical occurrence, unintended disease or injury or any untoward clinical signs (including an abnormal laboratory finding) in subjects, users or other persons whether or not related to the investigational medical device. Adverse event reports were elicited from the participants or resulted from the assessments at each study visit and recorded.
Arm/Group | CBL-101 Eye Drops | Vismed® Multi Eye Drops
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/38
Other Adverse Events (participants affected / at risk) | 2/45 | 1/38
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CBL-101 Eye Drops (N=45) | Vismed® Multi Eye Drops (N=38)
Eye irritation (Eye disorders) | 2 | 1

LIMITATIONS AND CAVEATS:
The participants were not masked to treatment as the compared products were provided in their original bottles to maintain their aseptic conditions but all the bottles were relabelled with no trade name. Labels and outer packaging were identical except for randomization number. Participants received sealed boxes and returned sealed boxes with instructions to keep the investigator masked.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor have at least 60 days to review any publication or presentation. The first release of results will involve all sites in this multicenter study.

DOCUMENTS (2):
  • Study Protocol (2018-06-06): https://cdn.clinicaltrials.gov/large-docs/02/NCT02975102/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-25): https://cdn.clinicaltrials.gov/large-docs/02/NCT02975102/SAP_001.pdf